CLINICAL TRIAL: NCT04280510
Title: Pathogenic Study of Adult Immune Enteropathies
Acronym: ENTEROPATH
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: C19-07; 2019-A01594-53 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-01-20; First posted 2020-02-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Celiac Disease; Autoimmune Enteropathy; Inflammatory Bowel Diseases
Keywords: Celiac Disease; Autoimmune enteropathy; Primary immunodeficiency; Intestinal lymphoma; Liver autoimmune diseases
MeSH Terms: conditions — Celiac Disease; Autoimmune enteropathy; Inflammatory Bowel Diseases; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Active coeliac patients: Patients with active coeliac disease
  Interventions: Genetic: Blood sample collection; gastrointestinal biopsy
- Treated coeliac patients: Patients with coeliac disease on gluten free diet
  Interventions: Genetic: Blood sample collection; gastrointestinal biopsy
- Sprue type I: Patients with refractory coeliac disease of type I
  Interventions: Genetic: Blood sample collection; gastrointestinal biopsy
- Sprue type II: Patients with refractory coeliac disease of type II
  Interventions: Genetic: Blood sample collection; gastrointestinal biopsy
- Intestinal Lymphoproliferations: Patients with intestinal lymphoproliferations
  Interventions: Genetic: Blood sample collection; gastrointestinal biopsy
- Non coeliac enteropathies: Patients with non coeliac immune-mediated enteropathy
  Interventions: Genetic: Blood sample collection; gastrointestinal biopsy
- Patients without neoplastic or inflammatory intestinal disease: Patients without neoplastic or inflammatory intestinal disease
  Interventions: Genetic: Blood sample collection; gastrointestinal biopsy

INTERVENTIONS:
Genetic: Blood sample collection; gastrointestinal biopsy — Targeted Next generation sequencing and whole exome sequencing Phenotyping of intestinal lymphocytes, single cell analyses, cytokines dosage...

SUMMARY:
The study focuses the mechanisms underlying the loss of intestinal homeostasis in celiac disease, refractory celiac disease and other immune diseases such as monogenic enteropathy, inflammatory bowel diseases or drug induced intestinal diseases. Mechanisms of transformation of lymphocytes leading to onset of lymphomatous complications of immune enteropathies will be investigated. Mechanisms of loss of hepatic lymphocytic homeostasis will also be assessed in liver associated diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* affiliated to social insurance
* signed informed consent

Exclusion Criteria:

* pregnancy
* under guardianship
* not able to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients planned to have blood specimens and possible upper and/or lower digestive endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2030-02-27 (Estimated); Study Completion 2033-02-27 (Estimated)

PRIMARY OUTCOMES:
Intestinal Lymphocytes count | Baseline
  Lymphocytes isolation
DNA sequencing | Baseline
  Targeted Next Generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Georgia MALAMUT, MD, PhD, Principal Investigator — APHP, Université de Paris (Université Paris Descartes)
Locations (4):
- France (4):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Saint Louis, Paris
  - Hôpital Cochin, Paris

IPD SHARING:
Plan to Share IPD: No